CLINICAL TRIAL: NCT06673433
Title: The Effect of Environmental Factors on the Macro-genome and Metabolism of Obese Patients.
Brief Title: The Effects of Environmental Factors on the Macro-genome and Metabolism of Obese Patients.
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 202-331-01
Record Dates: First submitted 2024-11-02; First posted 2024-11-04 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2024-11

CONDITIONS: Obesity and Overweight
Keywords: obesity; environment; air pollution; macrogenomics; metabolism
MeSH Terms: conditions — Obesity; Overweight | interventions — Adiposity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the obesity group: Patients diagnosed with obesity (body mass index (BMI) ≥ 28kg/m2)
  Interventions: Diagnostic Test: obesity
- the control group: Paticipants with nomal BMI （18.5 - 24 kg/m2)
  Interventions: Diagnostic Test: health

INTERVENTIONS:
Diagnostic Test: obesity — Patients diagnosed with obesity (BMI ≥ 28kg/m2)
  Groups: the obesity group
Diagnostic Test: health — the health control group include paticipants with nomal BMI
  Groups: the control group

SUMMARY:
The present study was designed to include obese patients diagnosed with obesity in the First Affiliated Hospital of Chongqing Medical University and a healthy control population. By analysing the relationship between metabolic parameters and macrogenomes in obesity, identifying key metabolic and macrogenomic differences between obese patients and healthy populations, and establishing the association between environmental factors and obesity-related metabolic disorders, the investigators will be able to provide new biomarkers and intervention targets for obesity prevention and treatment.

DETAILED DESCRIPTION:
Obese patients who attended the First Hospital of Chongqing Medical University and intended to undergo bariatric surgery were screened according to the inclusion and exclusion criteria. Patients' basic personal information and biological specimens including blood, faeces and urine were collected for metabolic and macro-genomic analyses. Air pollution exposure of the study subjects was collected by telephone follow-up. Metabolite profiles in blood and urine were analysed using liquid chromatography-mass spectrometry (LC-MS). Microbial community composition in faecal samples was analysed using 16S rRNA gene sequencing. Metabolic and macrogenomic differences between obese and control groups were compared using t-test or Mann-Whitney U-test. Logistic regression analyses were used to assess the independent effects of different environmental factors on metabolism and macrogenome. Identify key metabolites and microorganisms associated with obesity using Random Forest and Principal Component Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Obese patients with BMI ≥30kg/m2;
* Patients did not undergo surgical treatment before enrolment;
* Willing to participate in this study and sign the informed consent form;
* Complete clinical data.

Exclusion Criteria:

* Patients with systemic diseases such as severe cardiorespiratory insufficiency that affect the choice of treatment regimen;
* Pregnant or lactating women;
* Patients who are not suitable for enrolment as assessed by the investigator;
* Patients with incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study intend to include patients diagnosed with obesity in the First Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
BMI | BMI was examed when first join the study, whith through the whole study period, an average of 1 month.
  BMI = weight / height squared (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The Ethics Committee of this Clinical Centre does not allow the disclosure of patient information.